CLINICAL TRIAL: NCT00255320
Title: Experimental Headache Induced by Vasoactive Intestinal Polypeptide
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danish Headache Center (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: VIP-KASGlo2004
Record Dates: First submitted 2005-11-16; First posted 2005-11-18 (Estimated); Last update posted 2005-12-09 (Estimated); Status verified 2003-12

CONDITIONS: Healthy Volunteers, Headache, Migraine, Hemodynamics, VIP, SPECT, Ultrasound
Keywords: healthy volunteers, headache, migraine, hemodynamics, VIP, SPECT, ultrasound
MeSH Terms: conditions — Headache; Migraine Disorders

INTERVENTIONS:
Drug: VIP

SUMMARY:
We hypothesized that infusion of VIP may induce headache in healthy subjects and that VIP induced headache may be associated with dilatation of intra- and extracerebral blood vessels. To test this hypothesis, we performed a double blind placebo controlled crossover study in normal human volunteers and studied the effect on headache and cerebral as well as hemodynamic parameters.

DETAILED DESCRIPTION:
We hypothesized that infusion of VIP may induce headache in healthy subjects and that VIP induced headache may be associated with dilatation of intra- and extracerebral blood vessels. To test this hypothesis, we performed a double blind placebo controlled crossover study in normal human volunteers and studied the effect on headache and cerebral as well as hemodynamic parameters. In a double-blind, placebo-controlled, crossover design, the subjects were randomly allocated to receive 8 pmol/kg/min VIP or placebo (isotonic saline) over 25 min. Headache intensity, Mean velocity of blood flow in the middle cerebral artery (VmeanMCA), superfical temporal artery diameter, PetCO2, adverse events and vital signs were recorded at T-10, T0 and then every 10 min until 120 min after start of infusion. Single photon emission computerized tomography (SPECT) was performed at T-0, T20 and T60.

ELIGIBILITY:
Inclusion Criteria:

- healthy volunteers

Exclusion Criteria:

- migraine cerebrovascular disorders pregnancy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12
Dates: Start 2003-12; Study Completion 2004-06

PRIMARY OUTCOMES:
Headache intensity, Mean velocity of blood flow in the middle cerebral artery (VmeanMCA), superfical temporal artery diameter, PetCO2, adverse events and vital signs were recorded at T-10, T0 and then every 10 min until 120 min after start of infusion.

SECONDARY OUTCOMES:
All subjects were asked to complete a headache diary every hour until 10 h after the discharge. The diary included headache characteristics and accompanying symptoms according to the International Headache Society (IHS 2004)

CONTACTS AND LOCATIONS:
Overall Officials: Jakob Møller Hansen, MD, Study Chair — Danish Headache Center
Locations (1):
- Danish Headache Center , KAS Glostrup, Glostrup, Copenhagen, Denmark